CLINICAL TRIAL: NCT04402775
Title: Brachiocephalic Arteriovenous Fistulae: Two Different Techniques of Bloodless Surgery and Their Effect on Fistula Stenosis.
Acronym: ABAS
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Due to a low inclusion rate
Sponsor: HagaZiekenhuis (Other)
Responsible Party: Principal Investigator, M.J.C. de Kok, Medical student, HagaZiekenhuis
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: NL54827.098.15
Record Dates: First submitted 2016-04-16; First posted 2020-05-27 (Actual); Last update posted 2020-05-27 (Actual); Status verified 2020-05

CONDITIONS: Arteriovenous Fistula; Tourniquet; Stenosis
MeSH Terms: conditions — Arteriovenous Fistula; Constriction, Pathologic | interventions — Tourniquets

STUDY DESIGN:
Intervention Model Description: Patients eligible for the trial were randomly allocated to the tourniquet group (intervention) or vascular clamp group (control)
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Vascular clamps (No Intervention): Patients randomized to the use of vascular clamps to obtain a bloodless field during arteriovenous fistula surgery (standard protocol).
- Tourniquet (Experimental): Patients randomized to the use of a tourniquet to obtain a bloodless field during arteriovenous fistula surgery.
  Interventions: Other: Tourniquet

INTERVENTIONS:
Other: Tourniquet — A tourniquet will be used during surgery
  Arms: Tourniquet

SUMMARY:
Patients with a chronic kidney disease who opt for hemodialysis, needs a well-functioning hemodialysis access. The autologous arteriovenous fistula (AVF) is recognized as the golden standard of dialysis access. Unfortunately a great number of the AVFs fail to mature, and therefore cannot be used for dialysis. A significant stenosis is a major cause of nonmaturing AVFs. Remarkable are the stenoses that seem to develop in the venous outflow tract where the vascular clamp was located during surgery. The primary aim of this study was to compare bloodless surgery using vascular clamps and a tourniquet with respect to the development of hemodynamic or anatomical significant stenosis in patients with a brachiocephalic or radiocephalic AVF.

DETAILED DESCRIPTION:
Patients with a chronic kidney disease who opt for hemodialysis, needs a well-functioning hemodialysis access. The autologous arteriovenous fistula (AVF) is the golden standard of dialysis access. Unfortunately a great number of the AVFs fail to mature, and therefore cannot be used for dialysis. A significant stenosis is a major cause of nonmaturing AVFs.

Remarkable are the stenoses that seem to develop in the venous outflow tract where the vascular clamp was located during surgery. The primary aim of this study was to compare bloodless surgery using vascular clamps and a tourniquet with respect to the development of hemodynamic or anatomical significant stenosis in patients with a brachiocephalic or radiocephalic AVF.

ELIGIBILITY:
Inclusion Criteria:

* Mentally competent
* Written informed consent
* Age 18 years and older
* Indication for brachiocephalic AVF in HagaZiekenhuis
* Patient is able to complete the follow-up evaluation

Exclusion Criteria:

* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2016-04; Primary Completion 2018-07 (Actual); Study Completion 2018-07 (Actual)

PRIMARY OUTCOMES:
Stenosis postoperative (duplex ultrasonography) | 6 weeks
  Luminal vessel diameter

SECONDARY OUTCOMES:
Duration of surgery | During surgery
  Duration of surgery in minutes
AVF occlusion | Within 3 months after surgery
  AVF occlusion
Bleeding | Within 3 months after surgery
  Bleeding
Infection | Within 3 months after surgery
  Infection
Pseudoaneurysm | Within 3 months after surgery
  Pseudoaneurysm
Need for reintervention | 1 year postoperative
  Surgical or endovascular reintervention

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Biuckians A, Scott EC, Meier GH, Panneton JM, Glickman MH. The natural history of autologous fistulas as first-time dialysis access in the KDOQI era. J Vasc Surg. 2008 Feb;47(2):415-21; discussion 420-1. doi: 10.1016/j.jvs.2007.10.041. PMID 18241764
- [Background] Hodges TC, Fillinger MF, Zwolak RM, Walsh DB, Bech F, Cronenwett JL. Longitudinal comparison of dialysis access methods: risk factors for failure. J Vasc Surg. 1997 Dec;26(6):1009-19. doi: 10.1016/s0741-5214(97)70014-4. PMID 9423717
- [Background] Vascular Access 2006 Work Group. Clinical practice guidelines for vascular access. Am J Kidney Dis. 2006 Jul;48 Suppl 1:S176-247. doi: 10.1053/j.ajkd.2006.04.029. No abstract available. PMID 16813989
- [Background] Vascular Access Work Group. Clinical practice guidelines for vascular access. Am J Kidney Dis. 2006 Jul;48 Suppl 1:S248-73. doi: 10.1053/j.ajkd.2006.04.040. No abstract available. PMID 16813991
- [Background] Turmel-Rodrigues L, Mouton A, Birmele B, Billaux L, Ammar N, Grezard O, Hauss S, Pengloan J. Salvage of immature forearm fistulas for haemodialysis by interventional radiology. Nephrol Dial Transplant. 2001 Dec;16(12):2365-71. doi: 10.1093/ndt/16.12.2365. PMID 11733628
- [Background] Duijm LE, Overbosch EH, Liem YS, Planken RN, Tordoir JH, Cuypers PW, Douwes-Draaijer P, de Haan MW. Retrograde catheterization of haemodialysis fistulae and grafts: angiographic depiction of the entire vascular access tree and stenosis treatment. Nephrol Dial Transplant. 2009 Feb;24(2):539-47. doi: 10.1093/ndt/gfn526. Epub 2008 Sep 18. PMID 18802208
- [Background] Beathard GA, Arnold P, Jackson J, Litchfield T; Physician Operators Forum of RMS Lifeline. Aggressive treatment of early fistula failure. Kidney Int. 2003 Oct;64(4):1487-94. doi: 10.1046/j.1523-1755.2003.00210.x. PMID 12969170
- [Background] Turmel-Rodrigues L, Boutin JM, Camiade C, Brillet G, Fodil-Cherif M, Mouton A. Percutaneous dilation of the radial artery in nonmaturing autogenous radial-cephalic fistulas for haemodialysis. Nephrol Dial Transplant. 2009 Dec;24(12):3782-8. doi: 10.1093/ndt/gfp324. Epub 2009 Jul 1. PMID 19570886
- [Background] Grogan J, Castilla M, Lozanski L, Griffin A, Loth F, Bassiouny H. Frequency of critical stenosis in primary arteriovenous fistulae before hemodialysis access: should duplex ultrasound surveillance be the standard of care? J Vasc Surg. 2005 Jun;41(6):1000-6. doi: 10.1016/j.jvs.2005.02.019. PMID 15944600
- [Background] Richtlijn Shuntchirurgie, Nederlandse Vereniging voor Heelkunde. Utrecht; 2010.